CLINICAL TRIAL: NCT03223675
Title: Neurocognitive Impact and Dose-Effect Relationship of Hippocampal Avoidance During Whole Brain Radiotherapy Plus Simultaneous Integrated Boost - A Prospective Follow-up Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104-9176A3
Record Dates: First submitted 2017-06-22; First posted 2017-07-21 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Brain Metastasis; Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

ARMS (1):
- Hippocampus-sparing WBRT plus SIB (Experimental): All studied patients should undergo a computed tomography (CT) simulation scan encompassing the entire head region with 1.25-mm slice thickness using a thermoplastic mask for immobilization. To achieve conformal hippocampal sparing during the delivery of whole brain radiation (WBRT) and simultaneous integrated boost(s) (SIB), the technique of volumetric modulated arc therapy (VMAT) via Linac-based RapidArc®.In terms of dose prescription, a dose of 30 Gy in 12 fractions was prescribed to whole-brain planning target volume (PTV) containing the normal brain parenchyma; an simultaneous integrated boost up to 120 - 150% is attempted to irradiate the gross metastatic foci.
  Interventions: Radiation: hippocampal-sparing WBRT

INTERVENTIONS:
Radiation: hippocampal-sparing WBRT

SUMMARY:
For newly-diagnosed patients with brain metastasis, whole brain radiation therapy (WBRT) probably remains a common palliative management even for those with oligometastatic brain disease. However, WBRT-related late sequelae, particularly a decline in neurocognitive functions (NCFs), are a major concern. More importantly, in patients with limited brain metastases and a fair/good performance status, sparing the radiosensitive and vulnerable structures which are responsible for essential NCFs during the WBRT course is one of the reasonable strategies to postpone and prevent the development of WBRT-induced neurocognitive impairments. Actually, radiation-related neurocognitive dysfunction is usually characterized as a decline involving learning and memory, in which the extremely radiosensitive hippocampus indeed plays a critical role. In addition to the neurocognitive preservation by virtue of sparing the radiosensitive structures like the hippocampus, durable intracranial tumor control critically depends on an escalated radiotherapeutic dose level which is adequate enough to eradicate gross metastatic brain lesions. Therefore, in order to achieve both hippocampal sparing and simultaneous integrated boost(s) to gross metastatic foci, a specialized WBRT technique, hippocampal avoidance during WBRT plus simultaneous integrated boost (SIB) will be adopted in this prospective study. Moreover, the dose-effect relationship would be analyzed in order to explore the correlation between the equivalent uniform dose (EUD) irradiating the hippocampus and the neurocognitive change/decline after the above WBRT course measured by objective neurocognitive test tools. Newly-diagnosed cancer patients harboring 1-3 gross metastatic lesions but still in fair/good performance statuses are potentially eligible. All recruited patients should receive baseline functional brain MRI examination and baseline neurobehavioral assessment. Treatment planning will be designed via the technique of volumetric-modulated arc therapy (VMAT) to achieve both hippocampal avoidance and simultaneous integrated boost(s) to gross metastatic lesions. Except for the above regions for which conformal avoidance or SIB is attempted, the prescribed dose to the remaining brain parenchyma will be consistently 3000 cGy in 12 fractions. Accordingly, a battery of neuropsychological measures, which includes 7 standardized neuropsychological tests (e.g., executive functions, verbal and non-verbal memory, working memory, and psychomotor speed), is used to evaluate neurobehavioral functions for our registered patients. The primary outcome measure is delayed recall, as determined by the change/decline in verbal memory or non-verbal memory, from the baseline assessment to 4 months after the start of the WBRT course. This prospective cohort study aims to examine thoroughly the impact of a specialized WBRT technique, integrating both simultaneous integrated boost(s) delivered to gross metastatic foci and conformal hippocampal avoidance, on the status of NCF change/decline in patients with oligometastatic brain disease. It is anticipated that intracranial local control will be more sustainable and durable resulting from the escalated focal dose of SIBs. Ultimately, we also expect the dose-effect relationship will be clearly demonstrated after investigating the correlation between the hippocampal dosimetry and the status of NCF change/decline after receiving HA-WBRT plus SIB.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically-confirmed non-hematopoietic malignancy who are referred for therapeutic or prophylactic WBRT
* Good performance status no worse than Eastern Cooperative Group (ECOG) of 2 or a general status of Karnofsky Score (KPS) at least 70 %
* The number and extent of brain metastatic lesions should be no more than three metastatic foci with a greatest diameter no more than 3 cm

Exclusion Criteria:

* Patients with MRI-identified metastasis within 5 mm perihippocampally
* Patients with metastasis involving the brain stem
* Clinical suspicion of leptomeningeal spreading
* Patients with a solitary brain metastatic lesion which had been totally removed
* History of prior radiotherapy including stereotactic radiosurgery delivered to brain/head region for any reasons

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is delayed recall, as determined by the change/decline in verbal memory (WMS III- Word List score) from the baseline assessment to 4 months after the start of HS-WBRT. | 4 months after the start of HS-WBRT
  Neurocognitive assessment: including memory, executive functions, and psychomotor speed. This neurocognitive outcome was delayed recall, as determined by the change/decline in verbal memory [Wechsler Memory Scale - 3rd edition (WMS III) - Word List score] from the baseline assessment to 4 months after the start of the course of WBRT with hippocampus sparing (HS-WBRT). Additionally, the follow-up of neurocognitive assessment will also be administered at 12 months and up to 18 months after the start of HS-WBRT
The primary endpoint is delayed recall, as determined by the change/decline in non-verbal memory (WMS III- Visual Reproduction score) from the baseline assessment to 4 months after the start of HS-WBRT | 4 months after the start of HS-WBRT
  Neurocognitive assessment: including memory, executive functions, and psychomotor speed. This neurocognitive outcome was delayed recall, as determined by the change/decline in non-verbal memory (WMS III- Visual Reproduction score) from the baseline assessment to 4 months after the start of the course of WBRT with hippocampus sparing (HS-WBRT). Additionally, the follow-up of neurocognitive assessment will also be administered at 12 months and up to 18 months after the start of HS-WBRT.

SECONDARY OUTCOMES:
Overall survival time, indicated by the time from the date of recruitment to the date of expiring | up to 18 months
The time from the date of recruitment to that of intracranial progression/failure noted on brain MRI or CT | up to 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin SY, Tsan DL, Chuang CC, Yang CC, Pai PC, Wang CL, Wu YM, Lee CC, Lin CH, Wei KC, Chou WC. Oncological Outcomes After Hippocampus-Sparing Whole-Brain Radiotherapy in Cancer Patients With Newly Diagnosed Brain Oligometastases: A Single-Arm Prospective Observational Cohort Study in Taiwan. Front Oncol. 2022 Jan 12;11:784635. doi: 10.3389/fonc.2021.784635. eCollection 2021. PMID 35096584